CLINICAL TRIAL: NCT01464489
Title: Study of Intubation Time Required for Excellent Tracheal Intubation With Low Dose Rocuronium During Propofol Anaesthesia in Children With and Without Atropine
Brief Title: Intubation Time With Low Dose Rocuronium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AJIRB-MED-CT4-11-074
Record Dates: First submitted 2011-10-18; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Intubation; Difficult
Keywords: Intubation time; Atropine; Propofol anesthesia
MeSH Terms: interventions — Atropine; Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Experimental): Anaesthesia was induced with alfentanil 10 μg.kg-1, propofol 2.5 mg.kg-1 and rocuronium 0.3 mg.kg-1.And receive normal saline for control group
  Interventions: Drug: Atropine
- Atropine group (Active Comparator): Anaesthesia was induced with alfentanil 10 μg.kg-1, propofol 2.5 mg.kg-1 and rocuronium 0.3 mg.kg-1. And receive atropine (atropine sulfate) 10 μg.kg-1 for atropine group.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Atropine — Anaesthesia was induced with alfentanil 10 μg.kg-1, propofol 2.5 mg.kg-1 and rocuronium 0.3 mg.kg-1.
  Atropine(atropine sulphate) 10 μg.kg-1, intravenous injection during induction After 120 sec of atropine injection, record intubating condition
  Other Names: Atropine sulfate
  Arms: Control group
Drug: Normal saline — Anaesthesia was induced with alfentanil 10 μg.kg-1, propofol 2.5 mg.kg-1 and rocuronium 0.3 mg.kg-1 Normal saline intravenous injection during anesthetic induction After 120 sec of normal saline injection, record intubating condition
  Arms: Atropine group

SUMMARY:
The investigators hypothesized that increasing the cardiac output by use of atropine in children might result in a reduction of the intubation time needed to facilitate tracheal intubation.

DETAILED DESCRIPTION:
The investigators hypothesized that increasing the cardiac output by use of atropine in children might result in a reduction of the intubation time needed to facilitate tracheal intubation. Therefore, the purpose of this study was to determine TimeEI with a low dose of esmeron (rocuronium) (0.3 mg.kg-1) for achievement of successful tracheal intubation conditions during intravenous (i.v.) anaesthesia using propofol and alfentanil in children and to determine whether administration of i.v. atropine (atropine sulphate) (10 μg.kg-1) during anaesthesia induction reduced these times.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I,
* Tonsillectomy with adenoidectomy

Exclusion Criteria:

* Patients with known allergy to the drugs used in this study,
* A history of reactive airway disease and asthma,
* A neuromuscular disorder, an anticipated difficult airway, and
* Crying children on arrival in the operating theatre

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
intubation time | intubating condition at 120 seconds from rocuronium injection
  Tracheal intubation was attempted was predetermined according to the up-and-down method, starting with 120 s, in both groups. If intubation was successful (unsuccessful), the assigned intubation time was decreased (increased) by one interval for the next patients in that group, respectively. In this study, the investigators adopted 69, 83, 99, 120, 144, 173, and 208 s, since these intubation times have equal intervals (0.08) on a logarithmic scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD,PhD, Study Director — Ajou University School of Medicine
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Background] Stoddart PA, Mather SJ. Onset of neuromuscular blockade and intubating conditions one minute after the administration of rocuronium in children. Paediatr Anaesth. 1998;8(1):37-40. doi: 10.1046/j.1460-9592.1998.00719.x. PMID 9483596